CLINICAL TRIAL: NCT05791253
Title: Pain Management in Adults in Primary Intervention of the Mobile Emergency and Resuscitation Service of Pontoise
Brief Title: Pain Management in Primary Intervention of the Mobile Emergency and Resuscitation Service
Acronym: DOLSMUR
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD 1322
Record Dates: First submitted 2023-03-14; First posted 2023-03-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Pain
Keywords: Pain management; Emergency care; Mobile Emergency and Resuscitation Service
MeSH Terms: conditions — Pain; Agnosia | interventions — Pain Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pain management — Check whether pain management was carried out according to the recommendations of the French Society of Anaesthesia and Intensive Care (SFAR) and the French Society of Emergency Medicine (SFMU)

SUMMARY:
The aim of the study is to carry out an inventory of practices relating to the management of pain: its recognition, assessment and treatment.

DETAILED DESCRIPTION:
Pain is one of the most frequent reasons for seeking emergency care, with a prevalence of approximately 42% in pre-hospital care.

Pain management practices are defined by the French Society of Anaesthesia and Intensive Care (SFAR) and the French Society of Emergency Medicine (SFMU).

Pain must be systematically managed and treated. To do this, it is necessary to start by assessing the pain using self-assessment scales, the VAS (Visual Analogue Pain Scale) or the EN (Numerical Pain Scale) being the two validated scales.

Depending on the intensity of the pain, appropriate treatments should be prescribed:

* If EN < 6: level I or II analgesic
* If EN > 6: morphine titration Finally, after the treatment has been implemented, the pain must be re-evaluated using the same self-assessment scales in order to attest to the effectiveness of the treatment.

There is a lack of knowledge of the recommendations for pain management and assessment: 49% of SMUR doctors do not know the SFAR recommendations and only 17% define severe acute pain by a VAS or ENS greater than 6/10.

The aim of the study is to carry out an inventory of practices relating to the management of pain: its recognition, assessment and treatment and to check whether pain management was carried out according to the recommendations of the French Society of Anaesthesia and Intensive Care (SFAR) and the French Society of Emergency Medicine (SFMU).

ELIGIBILITY:
Inclusion Criteria :

* Patients over 18 years of age,
* Patient managed on primary intervention file between 01/11 and 30/11/2021, between 01/03 and 31/03/2022 or between 01/08 and 31/08/2022,
* Patient transferred to NOVO hospital (Pontoise, Beaumont-sur-Oise or Magny en Vexin site) for further medical care.

Exclusion Criteria :

* Patient in Cardiorespiratory Arrest (CRA),
* Patient in coma,
* Patient without applicant,
* Patient who has expressed his opposition to the collect of his data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received an intervention from the Mobile Emergency and Resuscitation Service (primary intervention) between 01/11 and 30/11/2021, between 01/03 and 31/03/2022 or between 01/08 and 31/08/2022.
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain management according to the recommendations of the SFAR and SFMU | At the end of the study, an average of one month
  The the recommendations of the SFAR and SFMU about Pain management is based on a composite criterion with the following items:
  * Pain recognition and assessment EN (Numerical scale)
  * Implementation of an adapted therapy (prescriptions) according to the pain scale scores
  * Re-evaluation of pain EN (Numerical scale)
  The evaluation of the objective is based on this composite criterion : for each item, the answer will be Yes or No. The outcom is validate if the answer of each item is yes.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Fancelli, Principal Investigator — Hospital NOVO - Pontoise site
Locations (1):
- Mobile Emergency and Resuscitation Unit - NOVO Hospital - Pontoise Site, Pontoise, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vivien B, Adnet F, Bounes V, Cheron G, Combes X, David JS, Diependaele JF, Eledjam JJ, Eon B, Fontaine JP, Freysz M, Michelet P, Orliaguet G, Puidupin A, Ricard-Hibon A, Riou B, Wiel E, de La Coussaye JE. [Sedation and analgesia in emergency structure. Reactualization 2010 of the Conference of Experts of Sfar of 1999]. Ann Fr Anesth Reanim. 2012 Apr;31(4):391-404. doi: 10.1016/j.annfar.2012.02.006. Epub 2012 Mar 28. No abstract available. French. PMID 22459942
- [Background] Galinski M, Ruscev M, Gonzalez G, Kavas J, Ameur L, Biens D, Lapostolle F, Adnet F. Prevalence and management of acute pain in prehospital emergency medicine. Prehosp Emerg Care. 2010 Jul-Sep;14(3):334-9. doi: 10.3109/10903121003760218. PMID 20507221
- [Background] Albrecht E, Taffe P, Yersin B, Schoettker P, Decosterd I, Hugli O. Undertreatment of acute pain (oligoanalgesia) and medical practice variation in prehospital analgesia of adult trauma patients: a 10 yr retrospective study. Br J Anaesth. 2013 Jan;110(1):96-106. doi: 10.1093/bja/aes355. Epub 2012 Oct 11. PMID 23059961
- [Background] Ricard-Hibon A, Chollet C, Saada S, Loridant B, Marty J. A quality control program for acute pain management in out-of-hospital critical care medicine. Ann Emerg Med. 1999 Dec;34(6):738-44. doi: 10.1016/s0196-0644(99)70099-5. PMID 10577403